CLINICAL TRIAL: NCT05752669
Title: The Role of Oxidative Stress and Mitochondrial TERT in the Progression and Therapeutic Resistance of Papillary Thyroid Cancer.
Brief Title: Oxidative Stress and Mitochondrial TERT in Papillary Thyroid Cancer.
Acronym: TEMPEST
Status: Completed | Type: Observational
Sponsor: Istituto Auxologico Italiano (Other)
Collaborators: University of Milan (Other)
Responsible Party: Sponsor
Other Study IDs: 05M902
Record Dates: First submitted 2023-02-21; First posted 2023-03-03 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Papillary Thyroid Cancer
MeSH Terms: conditions — Thyroid Cancer, Papillary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Oxidative stress (OS) could be involved in the progression of papillary thyroid cancer (PTC). Indeed, thyroid differentiation genes are silenced by a mechanism controlled by NOX4-derived OS. On the other hand, TERT contributes to mitochondrial OS protection, which could increase the resistance of cancer cells to therapeutic agents. The investigators aim to address the role of OS and mitochondrial TERT in the progression and therapeutic resistance of PTC. OS and TERT subcellular localization will be investigated in 150 PTCs and correlated to the genetic and expression profile of the tumors and to the clinical and prognostic features of the patients. Mechanisms implicated in TERT mitochondrial migration and the contribution of mitochondrial TERT to tumor progression will be investigated in cancer cell lines and primary cell cultures. This study will allow to identify OS as a marker of therapeutic resistance in PTC and will open new opportunities for the development of novel treatments targeting ROS generation/TERT nuclear export.

ELIGIBILITY:
Inclusion Criteria:

* Patients with papillary thyroid cancer
* Patients whose tumor and contralateral healthy tissues can be collected for the analyses

Exclusion Criteria:

* patients who did not provide consent
* patients lost at follow-up
* tissues not adequate for the analyses

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients operated for papillary thyroid cancer and followed by our Center of Excellence for the Diagnosis and Treatment of Thyroid Tumors.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2021-09-15 (Actual); Primary Completion 2025-05-31 (Actual); Study Completion 2025-05-31 (Actual)

PRIMARY OUTCOMES:
H202 generation (nmol/mg tissue) in papillary thyroid cancer and in corresponding normal tissues. | months 1-24
TERT mitochondrial localization (TERT/VDAC) in papillary thyroid tumors. | months 13-30
  TERT mitochondrial localization will be investigated by Western blot of mitochondrial fractions and normalized to VDAC protein expression.
Effect of exogenous oxidative stress (H2O2) and therapeutic agents (BRAF, MEK and Src kinase inhibitors) on TERT nuclear to mitochondrial translocation in thyroid cancer cell lines. | month 19-30
  TERT mitochondrial translocation will be measured by immunofluorescence.
Mitochondrial oxidative stress generation in cells lines treated with Src kinase inhibitors. | months 25-36
  Mitochondrial oxidative stress will be measured by immunofluorescence.
Proliferation in cells lines treated with Src kinase inhibitors. | months 25-36
  Proliferation will be measured by a colorimetric assay.
Apoptosis in cells lines treated with Src kinase inhibitors. | months 25-36
  Apoptosis will be measured by a luminometric assay.
Migration in cells lines treated with Src kinase inhibitors. | months 25-36
  Migration will be measured by wound healing assays.

SECONDARY OUTCOMES:
Genetic characterization of tumor tissues. | months 1-24
  Point mutations and fusions will be investigated in DNA and RNA, respectively,
Expression profile of tumor tissues. | months 1-24
  The expression level of 16 thyroid function genes will be investigated by a custom RNA sequencing panel.

CONTACTS AND LOCATIONS:
Overall Officials: Marina Muzza, PhD, Principal Investigator — Istituto Auxologico Italiano
Locations (1):
- Istituto Auxologico Italiano, Milan, Italy

REFERENCES:
- [Background] Muzza M, Colombo C, Cirello V, Perrino M, Vicentini L, Fugazzola L. Oxidative stress and the subcellular localization of the telomerase reverse transcriptase (TERT) in papillary thyroid cancer. Mol Cell Endocrinol. 2016 Aug 15;431:54-61. doi: 10.1016/j.mce.2016.05.005. Epub 2016 May 7. PMID 27164443
- [Background] Pesenti C, Muzza M, Colombo C, Proverbio MC, Fare C, Ferrero S, Miozzo M, Fugazzola L, Tabano S. MassARRAY-based simultaneous detection of hotspot somatic mutations and recurrent fusion genes in papillary thyroid carcinoma: the PTC-MA assay. Endocrine. 2018 Jul;61(1):36-41. doi: 10.1007/s12020-017-1483-2. Epub 2017 Dec 6. PMID 29214440
- [Background] Cancer Genome Atlas Research Network. Integrated genomic characterization of papillary thyroid carcinoma. Cell. 2014 Oct 23;159(3):676-90. doi: 10.1016/j.cell.2014.09.050. PMID 25417114
- [Background] Haugen BR, Alexander EK, Bible KC, Doherty GM, Mandel SJ, Nikiforov YE, Pacini F, Randolph GW, Sawka AM, Schlumberger M, Schuff KG, Sherman SI, Sosa JA, Steward DL, Tuttle RM, Wartofsky L. 2015 American Thyroid Association Management Guidelines for Adult Patients with Thyroid Nodules and Differentiated Thyroid Cancer: The American Thyroid Association Guidelines Task Force on Thyroid Nodules and Differentiated Thyroid Cancer. Thyroid. 2016 Jan;26(1):1-133. doi: 10.1089/thy.2015.0020. PMID 26462967
- [Background] Coperchini F, Croce L, Denegri M, Awwad O, Ngnitejeu ST, Muzza M, Capelli V, Latrofa F, Persani L, Chiovato L, Rotondi M. The BRAF-inhibitor PLX4720 inhibits CXCL8 secretion in BRAFV600E mutated and normal thyroid cells: a further anti-cancer effect of BRAF-inhibitors. Sci Rep. 2019 Mar 13;9(1):4390. doi: 10.1038/s41598-019-40818-w. PMID 30867499
- See also: PubMed ID: 27164443 — https://pubmed.ncbi.nlm.nih.gov/27164443/
- See also: PubMed ID: 29214440 — https://pubmed.ncbi.nlm.nih.gov/29214440/
- See also: PubMed ID: 25417114 — https://pubmed.ncbi.nlm.nih.gov/25417114/
- See also: PubMed ID: 26462967 — https://pubmed.ncbi.nlm.nih.gov/26462967/
- See also: PubMed ID: 30867499 — https://pubmed.ncbi.nlm.nih.gov/30867499/